CLINICAL TRIAL: NCT00001376
Title: Steroid Hormones, TH1/TH2 Cytokines and Reproductive Status
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940196; 94-AR-0196
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-07

CONDITIONS: Arthritis, Rheumatoid; Healthy; Pregnancy
Keywords: Androgens; Female; Immunology; Neuroendocrine Axis; Rheumatoid Arthritis; Postpartum; Pregnancy
MeSH Terms: conditions — Arthritis, Rheumatoid

SUMMARY:
This study is designed to evaluate blood Th1 and Th2 immunoregulatory cytokine production and hormonal levels associated with the third trimester of pregnancy and the postpartum state. Cytokine and hormone levels will be assessed in blood specimens obtained from healthy pregnant and postpartum females and compared to levels from premenopausal non-pregnant and non-postpartum females. Blood samples obtained at 30-36 weeks of gestation and 2-6 weeks postpartum will be the primary study points. Samples will also be obtained from pregnant, postpartum, and non-pregnant, non-postpartum, premenopausal female patients with rheumatoid arthritis. Additional data will be generated from samples from normal males, which will be compared with data from females.

We expect to find that pregnancy is associated with enhanced Th2 cytokine expression and that the postpartum state is associated with enhanced Th1 cytokine expression. We expect to see differences in cytokine expression between males and females as well. We seek to gather data supporting the view that distinct hormonal environments regulate these contrasting immunological states.

DETAILED DESCRIPTION:
This study is designed to evaluate blood Th1 and Th2 immunoregulatory cytokine production and hormonal levels associated with the third trimester of pregnancy and the postpartum state. Cytokine and hormone levels will be assessed in blood specimens obtained from healthy pregnant and postpartum females and compared to levels from premenopausal non-pregnant and non-postpartum females. Blood samples obtained at 30-36 weeks of gestation and 2-6 weeks postpartum will be the primary study points. Samples will also be obtained from pregnant, postpartum, and non-pregnant, non-postpartum, premenopausal female patients with rheumatoid arthritis. Additional data will be generated from samples from normal males, which will be compared with data from females.

We expect to find that pregnancy is associated with enhanced Th2 cytokine expression and that the postpartum state is associated with enhanced Th1 cytokine expression. We expect to see differences in cytokine expression between males and females as well. We seek to gather data supporting the view that distinct hormonal environments regulate these contrasting immunological states.

ELIGIBILITY:
No current medications or hormone therapy within the last 3 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 209
Dates: Start 1994-08; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bell SC, Billington WD. Major anti-paternal alloantibody induced by murine pregnancy is non-complement-fixing IgG1. Nature. 1980 Nov 27;288(5789):387-8. doi: 10.1038/288387a0. PMID 7432537
- [Background] Cadet P, Rady PL, Tyring SK, Yandell RB, Hughes TK. Interleukin-10 messenger ribonucleic acid in human placenta: implications of a role for interleukin-10 in fetal allograft protection. Am J Obstet Gynecol. 1995 Jul;173(1):25-9. doi: 10.1016/0002-9378(95)90164-7. PMID 7631699